CLINICAL TRIAL: NCT04496791
Title: Quality Control of CE-Certified Phonak Hearing Aids - 2020_26
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Sonova2020_26
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Root Canal Therapy; Hearing Aids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Successor of Phonak Audéo M-90 (Experimental): Phonak Hearing instrument (HI) with modified precalculation.
  Interventions: Device: RIC (Receiver in Canal) hearing aid/ hearing instrument (HI)
- Phonak Audéo M-90 (Active Comparator): Phonak Audéo M-90 is the most recent RIC device from Phonak which will be fitted to the participants individual hearing loss.
  Interventions: Device: RIC (Receiver in Canal) hearing aid/ hearing instrument (HI)

INTERVENTIONS:
Device: RIC (Receiver in Canal) hearing aid/ hearing instrument (HI) — HI is developed to support hearing impaired people in calm and complex situations and to be able to participate in communication

SUMMARY:
Phonak Hearing Devices pass through different development and study phases. At an early stage, feasibility studies are conducted to investigate new algorithms, features and functions in an isolated manner. If the benefit is proven, their performance is then investigated regarding interdependency between all available algorithms, features and functions running in parallel in a hearing aid (pivotal/pre-validation studies) and, resulting from the pre-validation studies, they get optimized. Prior to product launch, the Phonak Hearing Systems get reviewed by a final quality control in terms of clinical trials. This is a validation study, investigating improved algorithms, features, functions and wearing comfort. This will be a clinical investigation which will be conducted mono centric at Sonova AG Headquarters based in Stäfa (Switzerland).

DETAILED DESCRIPTION:
This study will investigate the combination of the features to determine if the audiological performance and quality of the new successor of the Marvel family shows an improved benefit over Phonak Audéo Marvel before going into the System Validation. Therefore this study will be a comparative study. The study will determine if hearing impaired users wearing the successor hearing aids, have better initial acceptance with the new precalculation, better sound quality and speech intelligibility, more clarity and loudness comfort in soft and loud environments compared to Phonak Marvel RIC (Receiver in channel) hearing aids. Another objective of the study is to compare the listening effort with the two different study devices.

ELIGIBILITY:
Inclusion Criteria:

* Hearing Loss range: N3-N4
* experienced hearing aid user
* willingness to wear behind the ear hearing aids
* Informed Consent as documented by signature

Exclusion Criteria:

* the audiogram is not in the fitting range of the intended hearing aid
* first time user
* limited mobility and not in the position to attend weekly appointments in Stäfa (Switzerland)
* participant is not able to describe experiences and hearing impressions
* allergies against the material of the hearing aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Rating of the sound quality for the new and the comparative HI | 4 weeks
  Subjective rating of the overall satisfaction for sound quality by questionnaires for the new HI and the old comparative HI (%). The participants rates after one week home trial. The home trial is randomized. The questionnaire includes rating scales for the satisfaction. The participant has to rate it in percentage (100% = very satisfy, 0% = very unsatisfy)

SECONDARY OUTCOMES:
Speech intelligibility in noisy situations (only test device) | 4 week
  Evaluating the speech intelligibility with the test device, using a speech in noise test, Oldenburger Satztest (OLSA) after the subject set the noise cancellation via an App on an individual limit. The results of the test are the word recognition score in SNR.
Speech intelligibility in quiet situations | 4 week
  Evaluating and comparing the speech intelligibility in a quiet test situation of the test device and the Marvel device. Using the "Reimtest nach Wallenberg und Kollmeier (WaKo ) (%).
Speech intelligibility in noisy situations | 4 weeks
  Evaluating and comparing the speech intelligibility in a noisy test situation of the test device and competitor. Using the OLSA (word recognition score)
Rating of sound quality | 1 week
  Subjective rating of the overall satisfaction for sound quality by questionnaires for the new HI and the old comparative HI (%). The participants rates after the First Fit. The questionnaire includes rating scales for the satisfaction. The participant has to rate it in percentage (100% = very satisfy, 0% = very unsatisfy)

CONTACTS AND LOCATIONS:
Locations (1):
- Sonova AG, Stäfa, Switzerland